CLINICAL TRIAL: NCT06429202
Title: Examination of the Relationship Between Body Perception and Self-Esteem Level and Quality of Life in Adolescent Idiopathic Scoliosis
Brief Title: The Relationship Between Body Perception and Self-Esteem Level and Quality of Life in Adolescent Idiopathic Scoliosis
Status: Not yet recruiting | Type: Observational
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Other Study IDs: Acetinkaya003
Record Dates: First submitted 2024-05-14; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Scoliosis; Adolescence; Self Esteem; Quality of Life
Keywords: idiopathic scoliosis; self esteem; body perception
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Scoliosis is a three-dimensional, multifactorial disease that becomes more prevalent in adolescents, disrupts the three-dimensional mechanism and posture of the vertebra, causes deterioration in the person's body perception and cosmetic perception, and also causes negative effects on social life and quality of life. Although idiopathic scoliosis is more common during adolescence, its cause is not yet known. It is divided into three subheadings according to the age of onset. These are respectively; It is classified as Juvenile Idiopathic Scoliosis (0-3 years), Infantile Idiopathic Scoliosis (4-10 years), Adolescent Idiopathic Scoliosis (10 years and above). The most common one is Adolescent Idiopathic Scoliosis. Its incidence in girls is 4 times higher than in boys. This study aimed to examine the effects of body image and self-esteem on quality of life in idiopathic adolescent scoliosis patients and to determine whether there is a difference between genders. Additionally, it will be examined what effect the duration of corset use has on these parameters.

DETAILED DESCRIPTION:
Scoliosis is a three-dimensional, multifactorial disease that becomes more prevalent in adolescents, disrupts the three-dimensional mechanism and posture of the vertebra, causes deterioration in the person's body perception and cosmetic perception, and also causes negative effects on social life and quality of life. Although idiopathic scoliosis is more common during adolescence, its cause is not yet known. It is divided into three subheadings according to the age of onset. These are respectively; It is classified as Juvenile Idiopathic Scoliosis (0-3 years), Infantile Idiopathic Scoliosis (4-10 years), Adolescent Idiopathic Scoliosis (10 years and above). The most common one is Adolescent Idiopathic Scoliosis. Its incidence in girls is 4 times higher than in boys. This study aimed to examine the effects of body image and self-esteem on quality of life in idiopathic adolescent scoliosis patients and to determine whether there is a difference between genders. Additionally, it will be examined what effect the duration of corset use has on these parameters. Thirty idiopathic adolescent scoliosis patients, boys and girls aged between 10 and 18, will be included in the study. Coopersmith Self-Esteem Inventory (CSEI) to evaluate body image, Walter Reed Visual Assessment Scale to evaluate body image, Scoliosis Research Society-22 Quality of Life Questionnaire to evaluate the level of quality of life, sociodemographic data form to obtain personal data, Statistical Package to analyze the data. for Social Science (SPSS) planned to use Windows version 22.0

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study and obtaining parental consent
* Being between the ages of 10-18
* Being diagnosed with idiopathic scoliosis
* Using a scoliosis brace for at least 3 months
* Being within the normal range in body mass index

Exclusion Criteria:

* Having previously undergone spine surgery, having any mental problems, having non-idiopathic scoliosis and orthopedic disease.
* Having a curve of less than 25 degrees

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 30 individuals between the ages of 10-18 diagnosed with Adolescent Idiopathic Scoliosis. As a general recommendation, Cohen states that if the d value is less than 0.2, the effect size can be defined as weak, if it is 0.5, it can be defined as medium, and if it is greater than 0.8, it can be defined as strong (Cohen, 1988). The minimum number of samples was calculated with the G*Power 3.1.9 program. Accordingly, the minimum number of samples to be included in the study for an effect size of 0.5, statistical power of 80% and margin of error of 0.05 was calculated as 29.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-10 (Estimated)

PRIMARY OUTCOMES:
Walter Reed Visual Assessment Scale | at baseline
  Walter Reed Visual Assessment Scale (WRGDS) is an evaluation scale created from visual figures. It was developed by Pineda et al. in 2006, for use in individuals with scoliosis, to measure how a person thinks about the deformity in their own body and how severe it is perceived.
Coopersmith Self-Esteem Inventory (CSEI) | at baseline
  It is a self-assessment scale developed by Stanley Coopersmith in 1967. This test aims to measure the individual's thoughts about himself and his general sense of self-esteem. The form consists of 58 questions and includes 50 self-esteem items and 8 lie items.
Scoliosis Research Society-22 Quality of Life Questionnaire | at baseline
  Scoliosis Research Society-22 is a 22-question quality of life scale specific to scoliosis. Developed by the Scoliosis Research Society, it has been translated into different languages and shown to be valid and reliable.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Çetinkaya, Principal Investigator — Halic University
Locations (1):
- Halic University, Istanbul, Eyupsultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No